CLINICAL TRIAL: NCT02607540
Title: Two-arm Phase III Trial Comparing Radiotherapy With Differentcycles of Cisplatin-5-fluorouracil for Esophageal Cancer
Brief Title: Different Cycles of Cisplatin-5-fluorouracil for the Chemoradiotherapy of Esophageal Squamous Cancer
Acronym: PFCRTESC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Henan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PF and esophageal cancer
Record Dates: First submitted 2015-11-16; First posted 2015-11-18 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Stage III Esophageal Squamous Cell Carcinoma; Stage II Esophageal Squamous Cell Carcinoma
Keywords: Chemoradiotherapy; Esophageal Squamous Cancer; Cisplatin-5-fluorouracil
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Two cycles PF-radiotherapy (Experimental): 2 cycles cisplatin-5-fluorouracil: cisplatin: 75mg/m2 d1，29；5-fluorouracil：750mg/m2 CIV24h d1-4，d29-32.
  radiotherapy： 50Gy，2 Gy/d，5d/w.
  Interventions: Other: 2 cycles cisplatin-5-fluorouracil; Radiation: Radiotherapy
- Four cycles PF-radiotherapy (Active Comparator): 4 cycles cisplatin-5-fluorouracil: cisplatin: 75mg/m2 d1，29, 57, 85；5-fluorouracil：750mg/m2 CIV24h d1-4，d29-32, d57-60, d85-88.
  radiotherapy： 50Gy，2 Gy/d，5d/w.
  Interventions: Other: 4 cycles cisplatin-5-fluorouracil; Radiation: Radiotherapy

INTERVENTIONS:
Other: 2 cycles cisplatin-5-fluorouracil — 2 cycles cisplatin-5-fluorouracil(PF 2 cycles): cisplatin: 75mg/m2 d1，29; 5-fluorouracil：750mg/m2 CIV24h d1-4，d29-32.
  Other Names: PF 2 cycles
  Arms: Two cycles PF-radiotherapy
Other: 4 cycles cisplatin-5-fluorouracil — 4 cycles cisplatin-5-fluoroura(PF 4 cycles): cilcisplatin: 75mg/m2 d1，29, 57, 85; 5-fluorouracil：750mg/m2 CIV24h d1-4，d29-32, d57-60, d85-88.
  Other Names: PF 4 cycles
  Arms: Four cycles PF-radiotherapy
Radiation: Radiotherapy — concurrent radiotherapy： 50Gy in total，2 Gy/d，5d/w，Until disease progression or unacceptable toxicity
  Other Names: Radiation Therapy

SUMMARY:
A two-arm Phase III trial was started in Oct. 2014. Definitive chemoradiotherapy with cisplatin plus 5-fluorouracil is the standard in Western countries in esophagus cancer. But in China because of its toxic reaction, most of patients stop the halfway.

The purpose of this study is to confirm the difference of 2 and 4 cycles of cisplatin plus 5-fluorouracil in the definitive chemoradiotherapy for esophagus squamous cell carcinoma. A total of 210 patients will be accrued from China within 2 years. The primary endpoint is overall survival and the secondary endpoints include progression-free survival, response rate, pathologic complete response rate and adverse events.

DETAILED DESCRIPTION:
We plan to recruit the patients who were pathologically confirmed with esophageal squamous cell carcinoma from the Oct 2014. The patients will be divided into two groups.Experimental group: Two cycles of cisplatin plus 5-fluorouracil concurrent radiotherapy.Control group:Four cycles of cisplatin plus 5-fluorouracil and concurrent radiotherapy.To evaluate the overall survival of the 2 group. Also observe the patient's progression-free survival, response rate, pathologic complete response rate and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* age 45-75years old
* Histologically proven squamous cell carcinoma of the esophagus the tumor was in T2-4N0-2M0
* The patients have not received the surgery or chemo-radiotherapy.
* Hb≥80g/L, absolute neutrophil count ≥1.5×109/L, Plt≥90×109/L,
* ALT、AST≤2.5*N,Cr≤1.5*N.
* performance status score 0-2

Exclusion Criteria:

* pregnant, lactating women
* Oxaliplatin or fluorouracil Allergy or metabolic disorders
* Radiotherapy contraindications
* History of organ transplantation
* Brain metastasis
* The peripheral nervous system disorders
* Severe infection
* Oral capecitabine who have difficulty with,such as dysphagia,The activities of digestive ulcer, Gastrointestinal bleeding
* Severe chronic diseases, such as, hepatopathy, nephropathy, respiratory disease,high blood pressure, diabetes.
* Other malignant tumor in recent 5 years.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2014-10; Primary Completion 2017-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
overall survival, OS | 2 years

SECONDARY OUTCOMES:
progression-free survival,PFS | 2 years
overall remission rate, ORR | 16 weeks
serious adverse event,SAE | 16 weeks
quality of life, Qol | 16 weeks
pathologic complete response rate | 16 weeks
disease control rate,DCR | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shegan Gao, Doctor, Study Chair — The First Affiliated Hospital of Henan University of Science and Technology; Tanyou Shan, Master, Study Director — The First Affiliated Hospital of Henan University of Science and Technology; Xiaoshan Feng, Doctor, Study Director — The First Affiliated Hospital of Henan University of Science and Technology; Jiachun Sun, Doctor, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Xinshuai Wang, Doctor, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Guoqiang Kong, Master, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Xiaozhi Yuan, Master, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Ruinuo Jia, Master, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Dan Zhou, Master, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Jing Ren, Master, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Ruina Yang, Master, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Wei Wang, Master, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Yongxuan Liu, Master, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Dan Wang, Master, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Shiyuan Song, Master, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Weijiao Yin, Master, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Yali Zhang, Master, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology
Locations (1):
- The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan, China

REFERENCES:
- [Background] Park JW, Kim JH, Choi EK, Lee SW, Yoon SM, Song SY, Lee YS, Kim SB, Park SI, Ahn SD. Prognosis of esophageal cancer patients with pathologic complete response after preoperative concurrent chemoradiotherapy. Int J Radiat Oncol Biol Phys. 2011 Nov 1;81(3):691-7. doi: 10.1016/j.ijrobp.2010.06.041. Epub 2010 Oct 1. PMID 20888705
- [Background] Minsky BD, Pajak TF, Ginsberg RJ, Pisansky TM, Martenson J, Komaki R, Okawara G, Rosenthal SA, Kelsen DP. INT 0123 (Radiation Therapy Oncology Group 94-05) phase III trial of combined-modality therapy for esophageal cancer: high-dose versus standard-dose radiation therapy. J Clin Oncol. 2002 Mar 1;20(5):1167-74. doi: 10.1200/JCO.2002.20.5.1167. PMID 11870157
- [Background] Ohtsu A, Boku N, Muro K, Chin K, Muto M, Yoshida S, Satake M, Ishikura S, Ogino T, Miyata Y, Seki S, Kaneko K, Nakamura A. Definitive chemoradiotherapy for T4 and/or M1 lymph node squamous cell carcinoma of the esophagus. J Clin Oncol. 1999 Sep;17(9):2915-21. doi: 10.1200/JCO.1999.17.9.2915. PMID 10561371
- [Background] Ishida K, Ando N, Yamamoto S, Ide H, Shinoda M. Phase II study of cisplatin and 5-fluorouracil with concurrent radiotherapy in advanced squamous cell carcinoma of the esophagus: a Japan Esophageal Oncology Group (JEOG)/Japan Clinical Oncology Group trial (JCOG9516). Jpn J Clin Oncol. 2004 Oct;34(10):615-9. doi: 10.1093/jjco/hyh107. PMID 15591460
- [Background] Hironaka S, Ohtsu A, Boku N, Muto M, Nagashima F, Saito H, Yoshida S, Nishimura M, Haruno M, Ishikura S, Ogino T, Yamamoto S, Ochiai A. Nonrandomized comparison between definitive chemoradiotherapy and radical surgery in patients with T(2-3)N(any) M(0) squamous cell carcinoma of the esophagus. Int J Radiat Oncol Biol Phys. 2003 Oct 1;57(2):425-33. doi: 10.1016/s0360-3016(03)00585-6. PMID 12957254
- [Background] Bedenne L, Michel P, Bouche O, Milan C, Mariette C, Conroy T, Pezet D, Roullet B, Seitz JF, Herr JP, Paillot B, Arveux P, Bonnetain F, Binquet C. Chemoradiation followed by surgery compared with chemoradiation alone in squamous cancer of the esophagus: FFCD 9102. J Clin Oncol. 2007 Apr 1;25(10):1160-8. doi: 10.1200/JCO.2005.04.7118. PMID 17401004
- [Background] Shapiro J, ten Kate FJ, van Hagen P, Biermann K, Wijnhoven BP, van Lanschot JJ. Residual esophageal cancer after neoadjuvant chemoradiotherapy frequently involves the mucosa and submucosa. Ann Surg. 2013 Nov;258(5):678-88; discussion 688-9. doi: 10.1097/SLA.0b013e3182a6191d. PMID 24096766
- [Background] Kato K, Nakajima TE, Ito Y, Katada C, Ishiyama H, Tokunaga SY, Tanaka M, Hironaka S, Hashimoto T, Ura T, Kodaira T, Yoshimura K. Phase II study of concurrent chemoradiotherapy at the dose of 50.4 Gy with elective nodal irradiation for Stage II-III esophageal carcinoma. Jpn J Clin Oncol. 2013 Jun;43(6):608-15. doi: 10.1093/jjco/hyt048. Epub 2013 Apr 12. PMID 23585687